CLINICAL TRIAL: NCT04959851
Title: Prospective, Non-Interventional, Observational Study in Patients With IBD Receiving IV or SC Vedolizumab Therapy to Observe Route of Administration Choices and Outcomes
Brief Title: A Study on How Vedolizumab is Given and the Outcomes for Adults With Inflammatory Bowel Disease (VARIETY-Belgium)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: MACS-2021-011101
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohns Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Inflammatory Bowel Disease (IBD): Participants diagnosed with moderately to severely active IBD (UC or CD) who are initiating or currently ongoing vedolizumab intravenous induction treatment or maintenance intravenous treatment in accordance with the current Summary of Product Characteristics (SmPC) along with the option to switch to vedolizumab subcutaneous (SC) treatment, will be observed prospectively for 24 months.

SUMMARY:
IBD consists of either ulcerative colitis or Crohn's disease.

The main aim of this study is to describe real-world treatment patterns in adults with moderate to severe ulcerative colitis or Crohn's disease when treated with vedolizumab. This will include how vedolizumab is given, which can either be an infusion through a vein (intravenous or IV), or an injection just under the skin (subcutaneous injection, or SC).

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with moderately to severely active IBD (UC or CD) who are initiating or currently ongoing induction or maintenance treatment with vedolizumab according to the current SmPC in the real world setting.

The study will enroll approximately 200 participants. The data will be collected prospectively and will be recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

• Participants with IBD

This multi-center study will be conducted in Belgium at specialized gastroenterology centers.

ELIGIBILITY:
Inclusion Criteria:

1. Has moderately to severely active IBD (UC or CD), initiating or ongoing IV induction treatment with vedolizumab in accordance with the current SmPC at baseline OR IBD participants receiving ongoing/maintenance IV vedolizumab treatment, with the option to switch to SC vedolizumab maintenance treatment.

Exclusion Criteria:

1. Prior history of intolerability, hypersensitivity, or other contraindications (active severe infections such as tuberculosis, sepsis, cytomegalovirus, listeriosis, and opportunistic infections such as Progressive Multifocal Leukoencephalopathy) to vedolizumab therapy as defined in the current SmPC.
2. Current or planned participation in an interventional clinical trial for CD or UC.
3. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderately to severely active UC or CD receiving vedolizumab treatment in accordance with the approved SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Persisting to Treatment With Vedolizumab IV Compared to Participants With Treatment Change Up to 12 Months | Baseline up to 12 months
Time to any Treatment Change | Baseline up to 24 months
Number of Participants With Reason for Treatment Change | Baseline up to 24 months
Number of Participants With Change in Vedolizumab Dosing Frequency | Baseline up to 24 months
Number of Participants Who Discontinued the Vedolizumab Treatment | Baseline up to 24 months
Number of Participants Who Changed to Another Treatment | Baseline up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- Belgium (10):
  - GZA St. Vincentius, Antwerp
  - UZA, Antwerp
  - Erasme, Brussels
  - ZOL, Genk
  - AZ St. Lucas, Ghent
  - CHR Citadelle, Liège
  - CHU Liège, Liège
  - CHC MontLégia, Liège
  - AZ Delta, Roeselaere
  - CHWAPI, Tournai

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60f13cd7f883ca001e82d337